CLINICAL TRIAL: NCT00747175
Title: A Randomized, Single-Blind, Placebo-Controlled, Single-Centre, Phase I Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics After Multiple Ascending Oral Doses of AZD1656 in T2DM Subjects
Brief Title: A Study to Evaluate Safety, Tolerability and P-Glucose After Multiple Ascending Oral Doses of AZD1656 in Type 2 Diabetes
Acronym: MAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Klas Malmberg, MD, PhD, Prof. Medical Science Director, Emerging Products, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: D1020C00002
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — AZD1656

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental): 3 (alt.4) gradually increasing repeated oral doses of AZD1656 given to 3 (alt.4) groups (6 on active and 2 on placebo in each group)
  Interventions: Drug: AZD1656
- 2 (Experimental): Oral dose of AZD1656 titrated during 3 days to a tolerable dose (15 on active and 5 on placebo)
  Interventions: Drug: AZD1656

INTERVENTIONS:
Drug: AZD1656 — Dose titration to 3 (alt 4) increasing dose-steps with oral suspension, 8 days treatment
  Arms: 1
Drug: AZD1656 — Dose titration of oral suspension to a tolerable dose, 1 month treatment
  Arms: 2

SUMMARY:
The purpose of this study is to assess safety and tolerability of AZD1656 after multiple repeated oral doses in patients with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Male or surgically sterile female of non-childbearing potential (post-menopausal, ie natural or induced menopause with last menstruation >1 year ago and LH and FSH in the post-menopausal range, and/or have undergone hysterectomy and/or bilateral oophorectomy
* Diagnosed diabetes Mellitus patients treated with diet and exercise alone or with up to two oral anti-diabetic drugs. Stable glycemic control indicated by no changed treatment within 3 months prior to enrollment
* HbA1c ≤10.5 % at screening (HbA1c value according to international DCCT standard)

Exclusion Criteria:

* Clinically significant illness or clinically relevant trauma, as judged by the investigator, within two weeks before the first administration of the IP
* History ischemic heart disease, stroke, transitorisk ischemic attack or symptomatic peripheral vascular disease
* Clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results. Positive test of Hepatitis B surface antigen, antibodies to HIV virus and antibodies to Hepatitis C virus

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Safety variables (AE, BP, pulse, plasma glucose, laboratory variables and ECG) | Blood samples taken repeatedly during 24 hours on study day sessions

SECONDARY OUTCOMES:
Pharmacokinetic variables | Blood samples taken repeatedly during 24 hours on study day sessions
Pharmacodynamic variables | Blood samples taken repeatedly during 24 hours on study day sessions

CONTACTS AND LOCATIONS:
Overall Officials: Klas Malmberg, MD, Phd, Prof, Study Director — AstraZeneca R&D Mölndal, SE-431 83 Mölndal, Sweden; Marcus Hompesch, MD, Principal Investigator — Profil Institute for Clinical Research, Inc.
Locations (1):
- Research Site, Chula Vista, California, United States